CLINICAL TRIAL: NCT05260424
Title: Predictors for Nasal Intermittent Positive Pressure Ventilation Failure for Premature Infants With Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E1-20-1250
Record Dates: First submitted 2021-10-20; First posted 2022-03-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome, Newborn; Premature
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-invasive ventilation failure: babies who will be intubated in the first 72 hours
  Interventions: Other: non-invasive ventilation
- non-invasive ventilation success: babies who will not intubated in the first 72 hours
  Interventions: Other: non-invasive ventilation

INTERVENTIONS:
Other: non-invasive ventilation — Babies who will have or won't have non-invasive ventilation failure in the first 72 hoursof life, will be compared.

SUMMARY:
Non-invasive respiratory support methods have been widely used in premature babies with respiratory distress syndrome (RDS) which has changed the basic management of premature babies in the early period. According to the 2019 European Guidelines on RDS management, early nasal CPAP is recommended as first-line therapy in infants <30 weeks of age who are at risk of RDS who do not require mechanical ventilation (MV). However, some of the premature babies have faced non-invasive ventilation failure. Remarkably, infants who experience non-invasive ventilation failure are at increased risk of death, pneumothorax, intraventricular hemorrhage, and bronchopulmonary dysplasia (BPD), among other morbidities. In non-invasive ventilation failure, although demographic factors such as small gestational age, low birth weight, and male gender play a role, it has been suggested that surfactant deficiency may also play an important role. The most frequently reported risk factor in predicting non-invasive failure in studies is the fraction of inspiring oxygen during the first hours of life. In addition, positive end-expiratory airway pressure (PEEP) required for patient stabilization was found to be a potential predictor. However, there are still limited data to predict non-invasive ventilation failure. "Which newborns are at high risk for non-invasive ventilation failure?" and "When should the surfactant be applied?". The study is a single-center, prospective study to evaluate prognostic factors, and most importantly to define the FiO2 threshold, which is an indicator of possible non-invasive ventilation failure in infants supported with nasal intermittent positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* <32 weeks preterm babies
* Those who have received nasal intermittent positive pressure ventilation

Exclusion Criteria:

* Babies born> 32 weeks
* Babies with congenital anomalies
* Babies who have intubated in the delivery room
* Babies whose parents refuse to participitate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Preterm babies < 32 weeks gestational age who have received nasal intermittent positive pressure ventilation.
Sampling Method: Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Risk of intubation in the first 72 hours in premature babies | 2 year
  To determine the risk of intubation in the first 72 hours of life in premature babies less than 32 weeks of gestation who have supported with nasal intermittent positive pressure ventilation

SECONDARY OUTCOMES:
To describe the incidence and early precursors of non-invasive ventilation failure. | 2 year
  Invasive, non-invasive ventilation and supplemental oxygen day time
Looking for early predictors, | 2 year
  Looking for early predictors, including combinations of breathed oxygen fraction (FiO2) and non-invasive ventilation level in early life
morbidity and mortality | 2 year
  To investigate the negative consequences of non-invasive ventilation failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dargaville PA, Aiyappan A, De Paoli AG, Dalton RG, Kuschel CA, Kamlin CO, Orsini F, Carlin JB, Davis PG. Continuous positive airway pressure failure in preterm infants: incidence, predictors and consequences. Neonatology. 2013;104(1):8-14. doi: 10.1159/000346460. Epub 2013 Apr 4. PMID 23595061
- [Background] Gulczynska E, Szczapa T, Hozejowski R, Borszewska-Kornacka MK, Rutkowska M. Fraction of Inspired Oxygen as a Predictor of CPAP Failure in Preterm Infants with Respiratory Distress Syndrome: A Prospective Multicenter Study. Neonatology. 2019;116(2):171-178. doi: 10.1159/000499674. Epub 2019 May 21. PMID 31112987
- [Background] Shi Y, Tang S, Zhao J, Shen J. A prospective, randomized, controlled study of NIPPV versus nCPAP in preterm and term infants with respiratory distress syndrome. Pediatr Pulmonol. 2014 Jul;49(7):673-8. doi: 10.1002/ppul.22883. Epub 2013 Sep 4. PMID 24039148